CLINICAL TRIAL: NCT02399631
Title: Implementation of an Enhanced Recovery Program After Laparoscopic Colon Cancer Surgery
Brief Title: Enhanced Recovery Program After Laparoscopic Colon Cancer Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Gyu-Seog Choi, Director, Head of colorectal cancer center, Principal Investigator, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNUHCRC005
Record Dates: First submitted 2015-03-09; First posted 2015-03-26 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Colon Cancer
Keywords: Perioperative treatment; Laparoscopic surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERAS group (Experimental): early recovery program with no preoperative mechanical bowel preparation, early diet initiation, and prevention of postoperative ileus after elective laparoscopic colon cancer surgery
  Interventions: Other: Enhanced recovery program
- Congrol group (No Intervention): Traditional, conventional perioperative treatment

INTERVENTIONS:
Other: Enhanced recovery program — Enhanced recovery program day-1: no mechanical bowel preparation, intake permit until 6 hrs before operation day0: operation, postoperative fluid therapy, antibiotics day1: liquid diet, early ambulation, removal of foley catheterization day2-3: soft diet day 4-5: discharge
  Arms: ERAS group

SUMMARY:
An enhanced recovery program has been developed to provide for colon cancer patients faster and more personalized postoperative treatment. Most of the previous studies have showed that the efficacy of the enhanced recovery program on both subjective and objective physical recovery of patients. However, such studies are rarely conducted in South Korea. The purpose of this study is to evaluate the feasibility and efficacy of a postoperative enhanced recovery program in patients who underwent laparoscopic colon cancer surgery at a tertiary hospital in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility rule of enrollment
* ECOG 0-2
* Pathologically diagnosed colon cancer
* Stage I-III
* No functional disturbance in liver, kidney, bone marrow
* Informed consent

Exclusion Criteria:

* Emergent operation
* Obstructive or perforated cancer
* Rectosigmoid or rectal cancer
* Synchronous tumor
* Uncontrolled psychiatric or neurologic problems
* Severe hepatic dysfunction (GOT, GPT ≥100IU/L)
* Renal dysfunction (Cr ≥2mg/dl)
* Recent MI, CVA, nitrate medication

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | 30 days post-operatively
  Duration of hospital stay from the date of operation to the date when a patient meets the following "discharge criteria".
  Discharge criteria:
  * Tolerance of consecutive 3 soft diet
  * Recovery of bowel function (without PONV)
  * No necessity of intravenous analgesics
  * Stable vital sign (afebrile)
Actual hospital stay | 30 days post-operatively

SECONDARY OUTCOMES:
Readmission rate | 30 days from time of surgery
30-day morbidity | 30 days from time of surgery
30-day mortality | 30 days from time of surgery
Quality of life | up to 30days from time of surgery
  EORTC QLQ-C30, before and after surgery
Nutritional status | up to 30days from time of surgery
  Body weight, body mass index, body composition, before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gyu-Seog Choi, MD, Study Chair — Kyunpook National Univercity Medical Center
Locations (1):
- Gyu seog Choi, Daegu, South Korea